CLINICAL TRIAL: NCT01420666
Title: Maxi-Analgesic OA Study: Multicentre, Double-blind, Placebo-controlled, Randomized, Parallel Group Comparison of the Effects of Maxigesic 325 With Acetaminophen or Ibuprofen on Patients With Pain From Osteoarthritis
Brief Title: Maxi-Analgesic Osteoarthritis (OA) Study
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was withdrawn for administrative reason
Sponsor: AFT Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFT-MX-7
Record Dates: First submitted 2011-08-16; First posted 2011-08-22 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Maxigesic 325 (Active Comparator): Maxigesic 325 (acetaminophen 325 mg + ibuprofen 97.5mg), three tablets four times a day, orally, with food
  Interventions: Drug: Maxigesic 325
- Acetaminophen (Active Comparator): Acetaminophen 325 mg, three tablets four times a day, orally, with food
  Interventions: Drug: Acetaminophen
- Ibuprofen (Active Comparator): ibuprofen 97.5mg, three tablets four times a day, orally, with food
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen 325 mg, three tablets four times a day, orally, with food
  Other Names: Paracetamol
  Arms: Acetaminophen
Drug: Maxigesic 325 — Maxigesic 325 (Acetaminophen 325 mg+ ibuprofen 97.5mg), three tablets four times a day, orally, with food
  Other Names: Actaminophen/paracetamol + ibuprofen
  Arms: Maxigesic 325
Drug: Ibuprofen — Ibuprofen 97.5mg, three tablets four times a day, orally, with food
  Arms: Ibuprofen
Drug: Placebo — placebo, three tablets four times a day, orally, with food
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether the analgesic effects of Maxigesic USA are greater than acetaminophen, ibuprofen or placebo in patients who have painful osteoarthritis of the hip or knee.

DETAILED DESCRIPTION:
Osteoarthritis is a significant and disabling disease in the developed world.

Published guidelines for medical management of osteoarthritis from expert groups, in general advocate acetaminophen as first line treatment. The European League Against Rheumatism (EULAR) guidelines (1)recommend acetaminophen should be first choice therapy in OA, and that NSAIDs should be reserved for those patients unresponsive to acetaminophen. The American College of Rheumatology Guidelines (2) recommend acetaminophen be considered as reasonable initial therapy in patients with mild to moderate OA pain and that NSAIDs be considered as an initial alternative in moderate to severe OA pain. The Canadian guidelines recommend acetaminophen for mild OA pain and NSAIDs for moderate to severe OA (3).

A Cochrane Review of acetaminophen in osteoarthritis concluded that NSAIDs were superior to acetaminophen for improving knee and hip pain in people with OA. However, it was noted that the size of the treatment effect was modest with NSAIDs appearing to be more effective in OA subjects with moderate-to-severe pain (4).

There are many situations in clinical practice where either acetaminophen alone or low dose ibuprofen is not sufficiently effective. In these cases the dose of acetaminophen cannot be increased to more than 4000mg/day due to toxicity concerns. In the case of ibuprofen the dose can be increased from 1200mg/day to 2400mg/day. However comparison of low dose ibuprofen with high dose showed gastrointestinal (GI) toxicity increased: the relative risk (RR) of GI complications increased from 1.6 (95% CI 0.8, 3.2) with low dose ibuprofen to 4.2 (95% CI 1.8, 9.8) with high dose ibuprofen (5). Ibuprofen is associated with a low risk of serious gastrointestinal complications, but this advantage is probably lost at doses above 1800 mg/day (6).

A simple combination treatment whereby both acetaminophen and ibuprofen can be taken together as one single tablet and at the same time each day would, if effective, have the advantage of increasing analgesia without having to raise the ibuprofen dose above 1200mg/day (1170mg if administered every 6 hours) and lose the improved safety profile associated with a lower dose of ibuprofen.

1. Pendleton A, Arden N, Dougados M, Doherty M, Bannwarth B, Bijlsma JW, et al. EULAR recommendations for the management of knee osteoarthritis: report of a task force of the Standing Committee for International Clinical Studies Including Therapeutic Trials (ESCISIT). Ann Rheum Dis. 2000;59(12):936-44.
2. Recommendations for the medical management of osteoarthritis of the hip and knee: 2000 update. American College of Rheumatology Subcommittee on Osteoarthritis Guidelines. Arthritis Rheum. 2000;43(9):1905-15.
3. Tannenbaum H, Peloso PM, Russell AS, Marlow B. An evidence-based approach to prescribing NSAIDs in the treatment of osteoarthritis and rheumatoid arthritis: The Second Canadian Consensus Conference. Can J Clin Pharmacol. 2000;7 Suppl A:4A-16A.
4. Towheed TE, Maxwell L, Judd MG, Catton M, Hochberg MC, Wells G. Acetaminophen for osteoarthritis. Cochrane Database Syst Rev. 2006(1):CD004257.
5. Henry D, Lim LLY, Garcia Rodriguez LA, Perez Gutthann S, Carson JL, Griffin M, et al. Variability in risk of gastrointestinal complications with individual non-steroidal anti-inflammatory drugs: Results of a collaborative meta-analysis. British Medical Journal. 1996;312 (7046):1563-6.
6. Henry D, McGettigan P. Epidemiology overview of gastrointestinal and renal toxicity of NSAIDs. Int J Clin Pract Suppl. 2003;Supplement.(135):43-9.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent before initiation of any study-related procedures.
* Have had symptoms of OA of the knee or hip for at least 6 months that has required analgesic medication.
* Have confirmed radiological evidence of OA.
* Be between 45 - 80 years of age inclusive, on the day of consent.
* In the opinion of a physician, require long term medication for treatment of painful OA.
* Have painful OA of the knee or hip with a pain score of at least 40 mm and no more than 80 mm on the WOMAC VAS pain scale at rest following a 3 - 7 day washout of existing analgesics.

Exclusion Criteria:

* Weigh less than 50 kg
* Rheumatoid arthritis or other inflammatory arthritis.
* Gout or recurrent episodes of pseudogout.
* Paget's disease.
* Articular fracture.
* Ochronosis.
* Acromegaly.
* Haemochromatosis.
* Wilson's Disease.
* Primary Osteochondromatosis.
* Heritable disorders (e.g. hypermobility).
* Have received or taken oral or parenteral corticosteroids within 2 months or intra-articular hyaluronic acid within 9 months.
* Has taken any single dose of an NSAID or acetaminophen within 12 hours prior to first dose of study drug
* Known to be pregnant or possibly pregnant
* Women of childbearing potential who, in the opinion of the investigator, are not using reliable contraception.
* Alcohol intake in excess of 14 units per week for females and 21 units per week for males.
* Have a history of drug abuse.
* Suffering from a neurological disorder relating to pain perception.
* In the opinion of the investigator, unable to understand the visual analogue pain score.
* Currently, or in the last 30 days, participating in a clinical trial involving another study drug.
* Suffering from any other diseases or conditions which, in the opinion of the investigator, means that it would not be in the patients best interests to participant in this study.
* Hypersensitivity to aspirin or other NSAID
* Hypersensitivity to acetaminophen
* Severe known haemopoietic, renal or hepatic disease, immunosuppression
* History of gastric ulceration, indigestion, stomach pain or GI bleeding or bleeding disorders
* Currently suffering from dehydration through diarrhoea and/or vomiting
* History of severe asthma defined as previous steroid treatment or hospital admission within the last 5 years.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
WOMAC pain intensity VAS | 13 weeks
  The difference between the week 13 average WOMAC pain intensity VAS and the baseline WOMAC VAS

SECONDARY OUTCOMES:
Time to peak analgesic effect | 13 weeks
  Time to peak analgesic effect using the WOMAC VAS pain intensity score (the average pain intensity score of that week).
Time-adjusted SPID | 13 weeks
  Time adjusted SPID obtained from the mean weekly WOMAC VAS pain intensity assessments over 13 weeks
Difference of WOMAC stiffness score | 13 weeks
  Difference between the week 13 WOMAC stiffness score and the baseline WOMAC stiffness score
Difference of WOMAC function score | 13 weeks
  Difference between the week 13 WOMAC function score and the baseline WOMAC function score
Time to rescue medication | 13 weeks
  Tie to rescue medication (oxycodone)
Safety | 13 weeks
  Adverse events (serious and non-serious) will be assessed during the blinded study period and up to 30 days after the last dose of study medication. Known NSAID adverse effects (i.e. GI ulceration, indigestion/stomach pain, bleeding, bronchospasm, water retention, renal failure, skin reactions and thromboembolic events) and known acetaminophen adverse effects (i.e. clinical evidence of hepatitis) will be compared between groups.
Time-adjusted WOMAC stiffness score | Over 13 weeks
  Time-adjusted WOMAC stiffness score over 13 weeks
Time-adjusted WOMAC function score | over 13 weeks
  Time-adjusted WOMAC function score over 13 weeks
Patient global assessment | 13 weeks
  A categorical global pain rating will be obtained weekly during the double blind treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: John Moodie, Doctor, Principal Investigator — Clinical Trial New Zealand Ltd, 32 Kahikatea Drive, Hamilton, New Zealand